CLINICAL TRIAL: NCT02155205
Title: Randomized, Double-blind, Placebo-controlled, Positive Controlled, 3-period, 6-sequence, Crossover Study to Define the Electrocardiogram Effects of a Single Dose of Telotristat Etiprate (LX1606) 1500 mg Compared With Placebo and Open Label Moxifloxacin in Healthy Subjects: A Thorough QT Study
Brief Title: A Thorough QT Study of Telotristat Etiprate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LX1606.1-105-NRM; LX1606.105 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: QT Interval
MeSH Terms: interventions — telotristat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telotristat etiprate (Experimental): Single dose of telotristat etiprate followed by a 7-day washout.
  Interventions: Drug: Telotristat etiprate
- Moxifloxacin (Active Comparator): Single dose of moxifloxacin followed by a 7-day washout.
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Single dose of placebo with a 7-day washout to follow.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telotristat etiprate — 1500 mg telotristat etiprate (six 250 mg tablets)
  Arms: Telotristat etiprate
Drug: Placebo — Matching placebo
  Arms: Placebo
Drug: Moxifloxacin — 400 mg moxifloxacin (one 400 mg tablet)
  Arms: Moxifloxacin

SUMMARY:
The purpose of this study is to demonstrate that telotristat etiprate does not differ from placebo in the mean change from Baseline QT interval corrected for heart rate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females ≥18 to ≤55 years of age (inclusive) at the time of Screening
* Body mass index ≥18 to ≤32 kg/m2 at Screening
* Vital signs (after at least 5 minutes resting in a supine position) at Screening which are within the following ranges: Systolic blood pressure 90 to 140 mm Hg, Diastolic blood pressure 50 to 90 mm Hg, heart rate 45 to 100 beats per minute (bpm)
* Clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], complete blood count, and urinalysis [UA]) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator
* Able to tolerate prolonged periods of quiet, motionless, supervised rest
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Able to comprehend and willing to sign an Informed Consent Form

Exclusion Criteria:

* Presence of clinically significant physical, laboratory, or ECG findings at Screening that, in the opinion of the Investigator or Sponsor, may interfere with any aspect of study conduct or interpretation of results
* >30 premature ventricular beats per hour on the Holter ECG monitoring at Day -1 of Period 1 (monitored at the clinic via telemetry)
* History of additional risk factors for torsade de pointes or the diagnosis or suggestion of a family history of short QT syndrome or long QT syndrome
* History of renal disease or significantly abnormal kidney function tests
* History of hepatic disease or significantly abnormal liver function tests
* History of any clinically significant psychiatric, renal, hepatic, pancreatic, cardiovascular, neurological, or gastrointestinal abnormality
* Concurrent conditions that could interfere with safety and tolerability measurements
* Positive hepatitis panel (including hepatitis B surface antigen and hepatitis C virus antibody) or positive human immunodeficiency virus antibody screens
* Use of tobacco, use of medications, or history of any disease or condition that might interfere with the conduct of the study in the opinion of the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline QT interval corrected for heart rate | Days 1-3

SECONDARY OUTCOMES:
Number of adverse events | 52 days
Plasma concentration of telotristat etiprate | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Suman Wason, MD, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Evansville, Indiana, United States